## Cover Page for Analysis Plan Document

Official Study Title: What makes people better at retrieving proper names?

NCT05550779

Document Date 9/5/24

Data analysis will be conducted using a two-way ANOVA for each of the TOT measures (TOTs/# familiar trials; TOTs/# known names TOTs/# unsuccessful retrievals) to determine significant main effects, interactions, and simple main effects between the variables. The proposed analysis will determine if there is a) a significant main effect of the manipulation on TOT rate, b) a significant main effect of age on TOT rate, and c) an interaction between mindfulness condition and age group on TOT rate. The two-way ANOVA will be conducted using SPSS (Version 28.0). First, main effects and interactions will be examined. If there is an interaction, simple main effects will be assessed using the Bonferroni adjustment.